CLINICAL TRIAL: NCT07309679
Title: The Effectivness of Two Herbal Mouth-washes Versus Chlorohexidine on Oral Health Among A Group of School Children
Brief Title: Effectiveness of Herbal vs Chlorhexidine Mouthwashes in Improving Oral Health in Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A04060922
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Plaque Score; Gingival Health; Streptococcus Mutans
MeSH Terms: interventions — chlorhexidine gluconate; Mouthwashes

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into three parallel groups, each receiving a different mouthwash:
  * Group I: Chlorhexidine (0.2%)
  * Group II: Pomegranate peel extract mouthwash
  * Group III: Neem extract mouthwash
  Each participant used only one type of mouthwash for the full 3-week study period. Comparisons were made between groups to evaluate differences in plaque index, gingival index, and salivary Streptococcus mutans levels.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chlorhexidine Mouthwash Group (Active Comparator): Participants used 0.2% chlorhexidine mouthwash . Each child rinsed with 5 ml twice daily (after breakfast and before bedtime) for 30 seconds under parental supervision for three weeks. This group served as the gold-standard control for evaluating the efficacy of herbal mouthwashes
  Interventions: Drug: Chlorhexidine Digluconate 0.2% Mouthwash
- Pomegranate Peel Extract Mouthwash Group (Experimental): Participants used a pomegranate peel extract (Punica granatum Linn.) mouthwash, prepared at Nanogate company. Each child rinsed with 5 ml twice daily (after breakfast and before bedtime) for 30 seconds under parental supervision for three weeks. The purpose was to evaluate its natural antimicrobial and anti-gingivitis effects compared to chlorhexidine.
  Interventions: Drug: Pomegranate Peel Extract Mouthwash
- Neem Extract Mouthwash Group (Experimental): Participants used a neem (Azadirachta indica) extract mouthwash, prepared at Nanogate company. Each child rinsed with 5 ml twice daily (after breakfast and before bedtime) for 30 seconds under parental supervision for three weeks. This group was designed to assess neem's potential antimicrobial and plaque-reducing effects relative to chlorhexidine and pomegranate mouthwashes.
  Interventions: Drug: Neem Extract Mouthwash

INTERVENTIONS:
Drug: Chlorhexidine Digluconate 0.2% Mouthwash — Commercially available 0.2% chlorhexidine digluconate mouthwash used as the gold standard control. Participants rinsed with 5 ml twice daily (after breakfast and before bedtime) for 30 seconds under parental supervision for three weeks. Used to compare the antimicrobial and anti-plaque effectiveness against herbal mouthwashes.
  Other Names: CHX; 0.2% CHX Mouthrinse
  Arms: Chlorhexidine Mouthwash Group
Drug: Pomegranate Peel Extract Mouthwash — Mouthwash containing pomegranate peel extract (Punica granatum Linn.), prepared at Nanogate company. Participants rinsed with 5 ml twice daily for 30 seconds for three weeks under parental supervision. The intervention aimed to evaluate pomegranate's natural anti-inflammatory and antimicrobial effects on plaque, gingivitis, and Streptococcus mutans levels
  Other Names: PPE Mouthwash; Punica granatum Mouthrinse
  Arms: Pomegranate Peel Extract Mouthwash Group
Drug: Neem Extract Mouthwash — Mouthwash containing neem extract (Azadirachta indica), prepared at Nanogate company. Participants rinsed with 5 ml twice daily for 30 seconds for three weeks under parental supervision. The intervention was designed to assess neem's antibacterial and plaque-reducing properties compared with chlorhexidine and pomegranate mouthwashes.
  Other Names: Azadirachta indica Mouthrinse; Neem Herbal Mouthwash
  Arms: Neem Extract Mouthwash Group

SUMMARY:
Dental plaque and gingivitis are common oral health problems among school children. Mechanical plaque control, such as tooth brushing, is essential but may be insufficient for maintaining optimal oral hygiene. Chlorhexidine mouthwash is considered the gold standard chemical plaque control agent; however, its long-term use is limited by side effects such as tooth staining and taste alteration. In recent years, herbal mouthwashes have gained attention as natural alternatives with fewer adverse effects.

This randomized, single-blinded clinical trial was conducted to evaluate the effectiveness of two herbal mouthwashes - pomegranate peel extract and neem extract - compared with 0.2% chlorhexidine mouthwash on oral health among school children aged 8-12 years in Mansoura City, Egypt. A total of 156 participants were divided into three groups based on the type of mouthwash used. Plaque index, gingival index, and salivary Streptococcus mutans levels were assessed at baseline and after three weeks.

The study aimed to determine whether herbal mouthwashes could provide comparable benefits to chlorhexidine in reducing plaque, gingivitis, and bacterial load, while offering better safety and compliance in children.

DETAILED DESCRIPTION:
Dental plaque is a biofilm composed of microbial communities that play a central role in the development of gingivitis and dental caries. Gingivitis is one of the most prevalent oral diseases among children, often resulting from the interaction between bacterial accumulation and host factors. Although mechanical plaque control through toothbrushing is the primary preventive measure, its effectiveness depends on manual skill and motivation, especially in children. Chemical plaque control using antimicrobial mouthwashes is therefore recommended as an adjunct.

Chlorhexidine (CHX) is considered the "gold standard" chemical agent for controlling plaque and gingival inflammation due to its broad-spectrum antimicrobial activity and substantivity. However, its long-term use is associated with side effects such as tooth staining, altered taste, and burning sensations, which can affect compliance. These limitations have encouraged the search for natural alternatives with fewer adverse effects and good acceptability, particularly for pediatric use.

This clinical trial evaluated the effectiveness of two herbal mouthwashes-pomegranate peel extract (Punica granatum Linn.) and neem extract (Azadirachta indica)-compared with chlorhexidine 0.2% mouthwash on oral health among school children in Mansoura City, Egypt. A randomized, single-blinded, parallel-group clinical trial design was adopted. A total of 156 children aged 8-12 years with a plaque index ≥1 were included and randomly assigned to one of three groups: Group I (chlorhexidine), Group II (pomegranate peel extract), and Group III (neem extract). Each participant used 5 ml of the assigned mouthwash twice daily for three weeks under parental supervision.

Plaque index (Silness and Löe), gingival index (Löe and Silness), and salivary Streptococcus mutans levels were measured at baseline and after three weeks. Compliance was monitored weekly. Data were analyzed using SPSS version 24 with a significance level of 0.05.

The study aimed to assess whether pomegranate peel and neem mouthwashes could produce plaque, gingival, and microbial reductions comparable to those of chlorhexidine, while providing improved safety and patient acceptability. Findings from this trial are expected to support the potential use of herbal mouthwashes as effective and natural alternatives for maintaining oral hygiene in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 12 years (common age group for gingivitis).
* Both male and female participants.
* Plaque Index ≥ 1 according to Silness and Löe index.
* Regular brushing habit (once per day).
* Parental consent obtained prior to participation.

Exclusion Criteria:

* Children with systemic diseases or conditions affecting salivary flow.
* Children with a history of antibiotic use within the last month before the study.
* Those with known allergy or intolerance to any mouthwash ingredients.
* Children currently using any other mouthwash or oral antiseptic.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Plaque Index (Silness & Löe) | baseline , 1 week , 2 weeks, 3 weeks
  Outcome measure: Mean change in Plaque Index score (Silness & Löe) from baseline to 3 weeks.
Gingival Index (Löe & Silness) | baseline , 1 week , 2 weeks, 3 weeks
  Mean change in Gingival Index score (Löe & Silness) from baseline to 3 weeks.
Salivary Streptococcus mutans Level | Baseline and 3 weeks after start of intervention
  Change in salivary Streptococcus mutans count (CFU/ml) from baseline to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rabab I Salama, professor, Principal Investigator — Faculty of Dentistry,Mansoura University
Locations (1):
- Faculty of Dentistry,Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared because the study involves children and contains sensitive health information.only aggregated results will be published.